CLINICAL TRIAL: NCT04701762
Title: Endotracheal Intubation Using Videolaryngoscopy Versus Conventional Direct Laryngoscopy: A Randomized Multiple Cross-over Cluster Trial
Brief Title: Endotracheal Intubation Using Videolaryngoscopy Versus Conventional Direct Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-1158
Record Dates: First submitted 2020-12-22; First posted 2021-01-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Intubation; Laryngoscopy
Keywords: Airway; Videolaryngoscope; Direct Laryngoscope

STUDY DESIGN:
Intervention Model Description: Cluster randomized multiple crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- videolaryngoscopy (Experimental): Initial intubation performed using GlideScope videolaryngoscope.
  Interventions: Device: GlideScope videolaryngoscope (Verathon, Bothell, Washington 98011)
- conventional direct laryngoscopy (Active Comparator): Initial intubation performed using direct laryngoscopy.
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: GlideScope videolaryngoscope (Verathon, Bothell, Washington 98011) — After confirming adequate muscle relaxation, initial laryngoscopy will be performed using GlideScope videolaryngoscope with an appropriately sized blade (usually size 3 or 4). The GlideScope (Verathon, Bothell, Washington 98011) is an FDA-cleared commercially available portable videolaryngoscope.
  Arms: videolaryngoscopy
Device: Direct laryngoscopy — After confirming adequate muscle relaxation, initial laryngoscopy will be performed using direct laryngoscopy with an appropriately sized Macintosh or Miller blade (usually size 3 or 4);
  Arms: conventional direct laryngoscopy

SUMMARY:
The investigators will evaluate the endotracheal intubation using video laryngoscopy versus conventional direct laryngoscopy on intubation success, quantified by the number of intubation attempts. The question is important because video laryngoscopes are more expensive than conventional direct laryngoscopes. The additional cost might be justified if video systems improve intubation success and reduce airway trauma. But if they do not, the extra cost would not be justified

DETAILED DESCRIPTION:
The investigators propose to enroll participants scheduled for elective or emergent cardiac, thoracic, or vascular surgery in the designated operating room suite who require endotracheal intubation for general anesthesia.

A cluster randomized multiple crossover design is used for this trial. The cardiac surgical suites will be divided into 2 sets of 11 operating rooms. Each set is treated as a unit and randomized to receive video or direct laryngoscopy in 1-week blocks, always with 1 set randomized to each approach. For analysis, each operating room within a set will be considered a separate cluster. Randomization will be conducted weekly on a 1:1 unstratified basis, using computer-generated codes maintained in a web-based system. Investigators access these codes a day before each new treatment block begins.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergent surgery requiring oral endotracheal intubation for general anesthesia.

Exclusion Criteria:

* The attending anesthesiologist prefers a specific approach for a particular patient
* Awake fiberoptic intubation is clinically indicated
* Insertion of double-lumen tube.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7736 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Ruetzler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ruetzler K, Bustamante S, Schmidt MT, Almonacid-Cardenas F, Duncan A, Bauer A, Turan A, Skubas NJ, Sessler DI; Collaborative VLS Trial Group. Video Laryngoscopy vs Direct Laryngoscopy for Endotracheal Intubation in the Operating Room: A Cluster Randomized Clinical Trial. JAMA. 2024 Apr 16;331(15):1279-1286. doi: 10.1001/jama.2024.0762. PMID 38497992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Protocol Enrollment (N = 7,736) is 172 less than the calculated total number of participants Started (N = 7908), because these patients were enrolled more than once and assigned to different clusters due to having multiple operations in designated operating rooms during the study.
Units Other Than Participants: surgical procedures
Groups:
- Cluster 1: Operating Suites 60 to 70: A cluster randomized multiple crossover design was used for this trial.
  The cardiac surgical suite was divided into 2 sets of 11 operating rooms each (cluster 1: operating suites 60 to 70, and cluster 2: operating suites 71 to 81). These sets are the clusters. All operations performed in these operating suites were assessed for eligibility. N= 172 patients were enrolled more than once and assigned to different clusters due to having multiple operations.
  Each week, one set of ORs was randomly assigned to video laryngoscopy, while the other set was assigned to direct laryngoscopy. At the beginning of each week, the randomization occurred again, so in the following week, the set of ORs that had video laryngoscopy might now be assigned to direct laryngoscopy, and vice versa. This randomization continues for 90 weeks, with each set of ORs potentially receiving a different intervention each week.
  For analysis, each operating room within a set was considered a separate cluster. Randomization was conducted weekly on a 1:1 unstratified basis, using computer-generated codes maintained in a web-based system. Investigators accessed these codes a day before each new treatment block began.
  N=1,945 patients with 1,995 operations were enrolled into cluster 1 during the 42 direct laryngoscopy periods (Randomization occurs weekly for 90 weeks). Additionally, 2,418 patients with 2,486 operations were enrolled in cluster 1 during the 48 video laryngoscopy periods.
- Cluster 2: Operating Suites 71 to 81: A total of 1,916 patients with 2,021 operations were enrolled into cluster 2 during the 48 direct laryngoscopy periods (Randomization occurs weekly for 90 weeks). Additionally, 1,828 patients with 1,927 operations were enrolled into cluster 2 during the 42 video laryngoscopy periods (Randomization occurs weekly for 90 weeks).
  In patients randomized to videolaryngoscopy, initial intubation was performed using GlideScope videolaryngoscope. GlideScope videolaryngoscope (Verathon, Bothell, WA 98011): After confirming adequate muscle relaxation, initial laryngoscopy will be performed using GlideScope videolaryngoscope with an appropriately sized blade (usually size 3 or 4). The GlideScope (Verathon, Bothell, WA 98011) is an FDA-cleared commercially available portable videolaryngoscope.
Period: Overall Study
Arm/Group | Cluster 1: Operating Suites 60 to 70 | Cluster 2: Operating Suites 71 to 81
Started | 4301; 4481 surgical procedures (N = 62 patients enrolled more than once and received both interventions due to having multiple operations in different periods.) | 3607; 3948 surgical procedures (N = 137 patients enrolled more than once and received both interventions due to having multiple operations in different periods.)
Direct Laryngoscopy | 1945; 1995 surgical procedures (In 42 direct laryngoscopy periods (Randomization occurs weekly for 90 weeks)) | 1916; 2021 surgical procedures (In 48 direct laryngoscopy periods (Randomization occurs weekly for 90 weeks))
Videolaryngoscopy | 2418; 2486 surgical procedures (In 48 video laryngoscopy periods (Randomization occurs weekly for 90 weeks).) | 1828; 1927 surgical procedures (In 42 video laryngoscopy periods (Randomization occurs weekly for 90 weeks).)
Completed | 4301; 4481 surgical procedures | 3607; 3948 surgical procedures
Not Completed | 0; 0 surgical procedures | 0; 0 surgical procedures

BASELINE CHARACTERISTICS:
Units Other Than Participants: surgical procedure
Groups:
- Videolaryngoscopy: Initial intubation performed using GlideScope videolaryngoscope.
  GlideScope videolaryngoscope (Verathon, Bothell, WA 98011): After confirming adequate muscle relaxation, initial laryngoscopy will be performed using GlideScope videolaryngoscope with an appropriately sized blade (usually size 3 or 4). The GlideScope (Verathon, Bothell, WA 98011) is an FDA-cleared commercially available portable videolaryngoscope.
- Total: Total of all reporting groups
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy | Total
Number analyzed (Participants) | 4196 | 3819 | 7736
Number analyzed (surgical procedure) | 4413 | 4016 | 8429
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (13) | 63 (14) | 63 (14)
Sex: Female, Male [Count of Units; unit: surgical procedure]
  Female | 2880 | 2599 | 5479
  Male | 1533 | 1417 | 2950
Race/Ethnicity, Customized [Count of Units; unit: surgical procedure]
  White/Caucasian | 3655 | 3293 | 6948
  Black | 411 | 410 | 821
  Other | 171 | 167 | 338
  Missing | 176 | 146 | 322
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: One missing in each group
  kg/m2
    number analyzed (surgical procedure) | 4412 | 4015 | 8427
    (all) | 29 (6.5) | 28 (6.0) | 28 (6.5)
Admission category [Count of Units; unit: surgical procedure]
  Elective | 3711 | 3424 | 7135
  Emergent | 702 | 592 | 1294
Surgery type [Count of Units; unit: surgical procedure]
  Cardiac | 3317 | 2934 | 6251
  Vascular | 559 | 560 | 1119
  Other | 474 | 453 | 927
  Thoracic | 63 | 69 | 132
ASA (American Society of Anesthesiologists) physical status [Count of Units; unit: surgical procedure]
  1 (Healthy) | 6 | 14 | 20
  2 (Mild systemic illness) | 74 | 94 | 168
  3 (Severe systemic illness) | 694 | 668 | 1362
  4 (Life-threatening systemic illness) | 3605 | 3211 | 6816
  5 (Not expected to survive without the operation) | 34 | 29 | 63
Level of first intubation clinician [Count of Units; unit: surgical procedure]
  CRNA | 1672 | 1611 | 3283
  Resident | 1357 | 1157 | 2514
  Fellow | 603 | 582 | 1185
  SRNA | 639 | 536 | 1175
  Attending anesthesiologist | 113 | 112 | 225
  Medical student | 29 | 18 | 47
Mallampati score [Count of Units; unit: surgical procedure] — To describe the relative size of the base of the tongue compared to the oropharyngeal opening in hopes of predicting the difficult airway.
  surgical procedure
    I (Soft palate, uvula, pillars visible) | 1078 | 1109 | 2187
    II (Soft palate, major part of uvula visible) | 2583 | 2406 | 4989
    III (Soft palate, base of uvula visible) | 660 | 453 | 1113
    IV (Only hard palate visible) | 64 | 24 | 88
    Missing | 28 | 24 | 52
History of difficult intubation within past 5 years [Count of Units; unit: surgical procedure] | 138 | 112 | 250

OUTCOME MEASURES:

1. Primary Outcome: The Number of Intubation Attempts With the Initial Laryngoscopy Instrument.
Description: Intubation attempts is defined as introduction and subsequent removal of a laryngoscope blade into the oral cavity whether or not the trachea was intubated.
Time Frame: From the start time of intubation to time of the end of surgery up to 24 hours.
Measure: Count of Units; unit: Surgical procedures
Units Other Than Participants: Surgical procedures
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy
Number analyzed (Participants) | 4196 | 3819
Number analyzed (Surgical procedures) | 4413 | 4016
Surgical procedures
  1 | 4336 | 3710
  2 | 70 | 277
  3 | 3 | 27
  >3 | 4 | 2
Statistical Analysis 1: Comparison: Videolaryngoscopy vs Conventional Direct Laryngoscopy; Test type: Superiority; p < 0.001, GLM cumulative logit GEE model; Odds Ratio (OR) = 0.20, 99.32% CI 2-sided [0.14 to 0.29]

2. Secondary Outcome: Intubation Failure
Description: Intubation failure is defined by the responsible clinician switching to an alternative laryngoscopy device for any reason at any time, or by more than 3 intubation attempts.
Time Frame: From the start time of intubation to time of the end of surgery.
Measure: Count of Units; unit: Surgical procedures
Units Other Than Participants: Surgical procedures
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy
Number analyzed (Participants) | 4196 | 3819
Number analyzed (Surgical procedures) | 4413 | 4016
Surgical procedures | 12 | 161
Statistical Analysis 1: Comparison: Videolaryngoscopy vs Conventional Direct Laryngoscopy; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Risk Ratio (RR) = 0.06, 99.32% CI 2-sided [0.03 to 0.14]

3. Secondary Outcome: Any Dental or Airway Injury
Description: Airway injury is defined as any bleeding or apparent injury to the lips, mouth, pharynx, vocal cords, or other airway structures recorded by the anesthesia team.
  Dental injury is defined as any apparent injury to the teeth as recorded by the anesthesia team.
Time Frame: From the start time of intubation to time of the end of surgery.
Measure: Count of Units; unit: Surgical procedures
Units Other Than Participants: Surgical procedures
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy
Number analyzed (Participants) | 4196 | 3819
Number analyzed (Surgical procedures) | 4413 | 4016
Surgical procedures | 41 | 42
Statistical Analysis 1: Comparison: Videolaryngoscopy vs Conventional Direct Laryngoscopy; Test type: Superiority; p = 0.53, GLM log-binomial model (log link); Risk Ratio (RR) = 0.87, 99.32% CI 2-sided [0.48 to 1.58]

4. Other Pre Specified Outcome: Maximum Mean Arterial Pressure
Description: Maximum mean arterial pressure (MAP) in the five minutes after intubation
Time Frame: In five minutes after intubation.
Population: N = 64 surgical procedures had missing MAP in the Videolaryngoscopy group; N = 39 procedures had missing MAP in the Direct laryngoscopy group.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Surgical procedures
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy
Number analyzed (Participants) | 4145 | 3784
Number analyzed (Surgical procedures) | 4349 | 3977
mmHg | 107 (24) | 105 (24)
Statistical Analysis 1: Comparison: Videolaryngoscopy vs Conventional Direct Laryngoscopy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [0.92 to 3.1]

5. Other Pre Specified Outcome: Maximum Heart Rate (HR)
Description: Maximum heart rate in the five minutes after intubation
Time Frame: In five minutes after intubation
Population: N = 26 procedures had missing HR in Videolaryngoscopy group; N = 17 procedures had missing HR in Direct laryngoscopy group.
Measure: Mean (Standard Deviation); unit: beats/min
Units Other Than Participants: Surgical procedures
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy
Number analyzed (Participants) | 4177 | 3805
Number analyzed (Surgical procedures) | 4387 | 3999
beats/min | 83 (18) | 83 (18)
Statistical Analysis 1: Comparison: Videolaryngoscopy vs Conventional Direct Laryngoscopy; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.34 to 1.2]

ADVERSE EVENTS:
Time Frame: From the start time of intubation to time of the end of surgery up to 24 hours.
Arm/Group | Videolaryngoscopy | Conventional Direct Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/4413 | 0/4016
Serious Adverse Events (participants affected / at risk) | 0/4413 | 0/4016
Other Adverse Events (participants affected / at risk) | 0/4413 | 0/4016

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT04701762/Prot_SAP_000.pdf